CLINICAL TRIAL: NCT01678638
Title: Timing of Inguinal Hernia Repair in Premature Infants: A Randomized Trial
Brief Title: Timing of Inguinal Hernia Repair in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Martin Blakely, Associate Professor of Pediatric Surgery and Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-225-01
Record Dates: First submitted 2012-08-30; First posted 2012-09-05 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Inguinal Hernia; Premature Birth of Newborn
Keywords: inguinal hernia; premature infants; anesthesia safety; neurodevelopmental outcome; preterm infants; neonatal prematurity
MeSH Terms: conditions — Hernia, Inguinal; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early inguinal hernia (IH) repair (Active Comparator): IH repair before NICU discharge
  Interventions: Procedure: IH repair before NICU discharge
- Late inguinal hernia (IH) repair (Active Comparator): IH repair as outpatient at approximately 55-60 weeks post-menstrual age
  Interventions: Procedure: IH repair at 55-60 weeks post-menstrual age

INTERVENTIONS:
Procedure: IH repair before NICU discharge — The IH repair is performed prior to NICU discharge (within 1-2 weeks of enrollment and randomization)
  Arms: Early inguinal hernia (IH) repair
Procedure: IH repair at 55-60 weeks post-menstrual age — The IH repair will be performed as an outpatient between approximately 55-60 weeks post-menstrual age.
  Arms: Late inguinal hernia (IH) repair

SUMMARY:
The purpose of this study is to determine whether early (before NICU discharge) or late (55-60 weeks post-menstrual age) inguinal hernia repair is safer for premature infants who have an inguinal hernia.

DETAILED DESCRIPTION:
This is a randomized clinical trial comparing early versus late repair in premature infants with an inguinal hernia (IH) to determine which approach may be safer. Safety in this trial is defined as the freedom from significant adverse events, a reduction in hospital days during the study period, and normal neurodevelopmental testing at 2 years. Costs of each treatment strategy are also important and are being evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Infant with estimated gestational age at birth of < 37 weeks, 0 days
* In a NICU at participating site
* Diagnosed with an IH per the pediatric surgery team
* Parents and providers willing to randomize the infant

Exclusion Criteria:

* Infant is undergoing another operative procedure and IH repair is planned as a secondary procedure (e.g. fundoplication or G tube is planned, and IH repair is considered a secondary procedure)
* Known major congenital anomaly that impacts neurodevelopmental outcome or chromosomal abnormality
* Family unable to return for follow up and later IH repair; or likely unable to monitor IH as outpatient

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 338 (Actual)
Dates: Start 2013-06; Primary Completion 2023-04 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Significant adverse event (SAE) rate | 9 months beyond NICU discharge
  Specific significant adverse events that are either treatment related or hernia related have been defined a priori and will be assessed in both groups from randomization until 9 months after NICU discharge.
Number of hospital days | From randomization until 9 months post NICU discharge
  Total number of hospital days

SECONDARY OUTCOMES:
Hospital costs | Enrollment through 9 months after NICU discharge
  Departmental level costs at each participating institution will be determined for care that occurs from randomization until 9 months post NICU discharge.
Bayley Scales of Infant Development, 3rd Edition | 22-26 months corrected age
  Mean BSID scores; primarily cognitive domain

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Blakely, MD, MS, Principal Investigator — Vanderbilt University Medical Center; Jon E Tyson, MD, MPH, Principal Investigator — University of Texas Health Science Center at Houston; Children's Memorial Hermann Hospital
Locations (40):
- United States (40):
  - University of Alabama at Birmingham School of Medicine; Children's Hospital of Alabama, Birmingham, Alabama
  - University of Arkansas for Medical Sciences; Arkansas Children's Hospital, Little Rock, Arkansas
  - Southern California Permanente Group, Los Angeles, California
  - University of California, Los Angeles David Geffen School of Medicine; Mattel Children's & LA Biomed, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Naval Medical Center San Diego, San Diego, California
  - UCSD Rady Children's Hospital, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - UF Health Shands Children's Hospital, Gainesville, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota Medical School; Amplatz Children's Hospital, Minneapolis, Minnesota
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine in St. Louis; St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital & Medical Center of Omaha, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - Oishei Children's Hospital of Buffalo, Buffalo, New York
  - Columbia University Irving Medical Center, New York, New York
  - Cohen Children's Medical Center, Queens, New York
  - Duke University Medical Center; Duke Children's Hospital and Health Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Ohio State University College of Medicine; Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - OHSU Doernbecher Children's Hospital, Portland, Oregon
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital at Erlanger UT Chattanooga, Chattanooga, Tennessee
  - University of Tennessee Health Science Center; Le Bonheur Children's Hospital, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas, Southwestern Medical Center; Children's Medical Center, Dallas, Texas
  - Baylor College of Medicine; Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston; Children's Memorial Hermann Hospital, Houston, Texas
  - Primary Children's Hospital University of Utah, Salt Lake City, Utah
  - UVA Children's Hospital, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center; Children's Hospital of Richmond, Richmond, Virginia
  - University of Washington School of Medicine; Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin; Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] HIP Trial Investigators; Blakely ML, Krzyzaniak A, Dassinger MS, Pedroza C, Weitkamp JH, Gosain A, Cotten M, Hintz SR, Rice H, Courtney SE, Lally KP, Ambalavanan N, Bendel CM, Bui KCT, Calkins C, Chandler NM, Dasgupta R, Davis JM, Deans K, DeUgarte DA, Gander J, Jackson CA, Keszler M, Kling K, Fenton SJ, Fisher KA, Hartman T, Huang EY, Islam S, Koch F, Lainwala S, Lesher A, Lopez M, Misra M, Overbey J, Poindexter B, Russell R, Stylianos S, Tamura DY, Yoder BA, Lucas D, Shaul D, Ham PB 3rd, Fitzpatrick C, Calkins K, Garrison A, de la Cruz D, Abdessalam S, Kvasnovsky C, Segura BJ, Shilyansky J, Smith LM, Tyson JE. Effect of Early vs Late Inguinal Hernia Repair on Serious Adverse Event Rates in Preterm Infants: A Randomized Clinical Trial. JAMA. 2024 Mar 26;331(12):1035-1044. doi: 10.1001/jama.2024.2302. PMID 38530261